CLINICAL TRIAL: NCT05065190
Title: A Double Blind, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of Nintedanib Over 52 Weeks in Chinese Patients With Chronic Fibrosing ILDs With a Progressive Phenotype
Brief Title: A Study to Test How Well a Medicine Called Nintedanib Helps People in China With Progressive Lung Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1199-0434
Record Dates: First submitted 2021-09-30; First posted 2021-10-01 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 mg Nintedanib (Experimental): A soft gelatin capsule of 150 mg Nintedanib was administered orally twice daily (bid) in Chinese patients with chronic fibrosing ILD with progressive phenotype with over 52 weeks. Dose could be reduced to 100 mg bid to manage adverse events.
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): A soft gelatin capsule of placebo matching in size, weight, colour and shape to 150 milligram (mg) or 100 mg soft gelatin capsule of Nintedanib, was administered orally twice daily (bid) in Chinese patients with chronic fibrosing Interstitial Lung Disease (ILD) with progressive phenotype with over 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Soft gelatin capsule
  Arms: 150 mg Nintedanib
Drug: Placebo — Soft gelatin capsule
  Arms: Placebo

SUMMARY:
This study in China is open to people with progressive lung fibrosis (chronic fibrosing ILDs with progressive phenotype) who are at least 18 years old. The purpose of this study is to find out whether a medicine called nintedanib helps people with progressive lung fibrosis.

Participants are put into 2 groups randomly, which means by chance. 1 group gets nintedanib as capsules twice a day. The other group gets placebo as capsules twice a day. Placebo capsules look like nintedanib capsules but do not contain any medicine.

Participants are in the study for about 1 year. During this time, they visit the study site about 10 times. At some visits, participants perform a lung function test. The doctors check whether study treatment can slow down the loss of lung function. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent consistent with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local laws signed prior to entry into the study (and prior to any study procedure including shipment of High-Resolution Computed Tomography (HRCT) to reviewer.
* Male or female patients aged ≥ 18 years at Visit 1.
* Patients with physician diagnosed Interstitial Lung Disease (ILD) who fulfil at least one of the following criteria for Progressive Phenotype within 24 months of screening visit (Visit 1) despite treatment with unapproved medications used in clinical practice to treat ILD, as assessed by the investigator:

  * Clinically significant decline in Forced Vital Capacity (FVC) % predicted based on a relative decline of ≥10%
  * Marginal decline in FVC % predicted based on a relative decline of ≥5-<10% combined with worsening of respiratory symptoms
  * Marginal decline in FVC % predicted based on a relative decline of ≥5-<10% combined with increasing extent of fibrotic changes on chest imaging
  * Worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest imaging [Note: Changes attributable to comorbidities e.g. infection, heart failure must be excluded. Unapproved medications used in the clinical practice to treat ILD include but are not limited to corticosteroid, azathioprine, mycophenolate mofetil (MMF), n-Acetylcysteine (NAC), rituximab, cyclophosphamide, cyclosporine, tacrolimus].
* Fibrosing lung disease on HRCT, defined as reticular abnormality with traction bronchiectasis with or without honeycombing, with disease extent of >10%, performed within 12 months of Visit 1 as confirmed by central readers.
* For patients with underlying Connective Tissue Disease (CTD): stable CTD as defined by no initiation of new therapy or withdrawal of therapy for CTD within 6 weeks prior to Visit 1.
* FVC ≥ 45% predicted at Visit 2.

Exclusion Criteria:

* Aspartate Aminotransferase (AST) and / or Alanine Aminotransferase (ALT) > 1.5 x Upper Level of Normal (ULN) at Visit 1
* Bilirubin > 1.5 x ULN at Visit 1
* Creatinine clearance <30 milliliter (mL)/minute (min) calculated by Cockcroft-Gault formula at Visit 1.

[Note: Laboratory parameters from Visit 1 have to satisfy the laboratory threshold values as shown above. Visit 2 laboratory results will be available only after randomization. In case at Visit 2 the results do no longer satisfy the entry criteria, the Investigator has to decide whether it is justified that the patient remains on study drug. The justification for decision needs to be documented. Laboratory parameters that are found to be abnormal at Visit 1 are allowed to be re-tested (once) if it is thought to be a measurement error (i.e. there was no abnormal result of this test in the recent history of the patient and there is no related clinical sign) or the result of a temporary and reversible medical condition, once that condition is resolved].

* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment).
* Previous treatment with nintedanib or pirfenidone.
* Other investigational therapy received within 1 month or 6 half-lives (whichever was greater) prior to screening visit (Visit 1).
* Use of any of the following medications for the treatment of Interstitial Lung Disease (ILD): azathioprine (AZA), cyclosporine, Mycophenolate Mofetil (MMF), tacrolimus, oral corticosteroids (OCS) >20mg/day and the combination of OCS+AZA+ n-Acetylcysteine (NAC) within 4 weeks of Visit 2, cyclophosphamide within 8 weeks of Visit 2, rituximab within 6 months of Visit 2.

Note: Patients whose Regulatory Authority (RA)/Connective Tissue Disease (CTD) is managed by these medications should not be considered for participation in the current study unless change in RA/CTD medication is medically indicated.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - China-Japan Friendship Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - West China Hospital, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Med College, Wenzhou
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - General Hospital of Ningxia Medical University, Yinchuan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A double blind, randomized, placebo-controlled trial to generate additional data on the efficacy of 150 mg bid nintedanib in Chinese patients with Chronic Fibrosing Interstitial Lung Disease (ILD) with a progressive phenotype compared with placebo over 52 weeks.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | 150 mg Nintedanib
Started | 27 | 54
Completed (= Not prematurely discontinued from trial medication before 52 weeks) | 20 | 32
Not Completed | 7 | 22
Not completed — Other than listed | 2 | 12
Not completed — Lack of Efficacy | 4 | 0
Not completed — Adverse Event | 1 | 10

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who were randomized to a treatment group and received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg Nintedanib | Total
Number analyzed (Participants) | 27 | 54 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (8.4) | 63.8 (8.4) | 64.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 28 | 44
  Male | 11 | 26 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 54 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 54 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC) Over 52 Weeks Expressed in Milliliter (mL)
Description: Annual rate of decline in FVC over 52 weeks expressed in milliliter (mL). The main analysis used a restricted maximum likelihood (REML)-based approach with a random slope and intercept model. The analysis included the fixed, categorical effects of treatment, high resolution computed tomography (HRCT) pattern at baseline, fixed continuous effects of time and baseline FVC as well as the treatment-by-time and baseline-by-time interactions. Random effects were included for the patient response for both time and intercept.
  For patients who prematurely discontinued study treatment, data collected at follow-up visit and visits after treatment discontinuation was included in the analysis.
Time Frame: From baseline up to Week 52.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Milliliter/year
Arm/Group | Placebo | 150 mg Nintedanib
Number analyzed (Participants) | 27 | 54
Milliliter/year | -191.89 [-313.15 to -70.63] | -85.32 [-176.40 to 5.76]
Statistical Analysis 1: Comparison: Placebo vs 150 mg Nintedanib; Test type: Other; Adjusted difference = 106.57, 95% CI 2-sided [-47.13 to 260.28], Standard Error of Mean 76.84 — Adjusted difference between treatment groups was based on a random slope and intercept model with fixed effects for treatment, HRCT pattern, and baseline FVC [mL], and including treatment-by-time and baseline-by-time interactions

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and other adverse events: From first drug intake until end of trial visit, plus 7 days of residual effect period, up to 53 weeks.
Description: Treated Set (TS): All patients who were randomized to a treatment group and received at least one dose of study medication.
Arm/Group | Placebo | 150 mg Nintedanib
All-Cause Mortality (participants affected / at risk) | 3/27 | 6/54
Serious Adverse Events (participants affected / at risk) | 12/27 | 20/54
Other Adverse Events (participants affected / at risk) | 23/27 | 51/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | 150 mg Nintedanib (N=54)
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 2
Complicated appendicitis (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Myocardial necrosis marker increased (Investigations) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | 150 mg Nintedanib (N=54)
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 19
Nausea (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 7
Chest pain (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 4
Pyrexia (General disorders) | 2 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 12
Liver injury (Hepatobiliary disorders) | 0 | 3
COVID-19 (Infections and infestations) | 7 | 14
Influenza (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 7
Urinary tract infection (Infections and infestations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 10
Aspartate aminotransferase increased (Investigations) | 2 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 5
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 1 | 10
Lymphocyte percentage decreased (Investigations) | 0 | 3
Neutrophil percentage increased (Investigations) | 0 | 4
Weight decreased (Investigations) | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05065190/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT05065190/SAP_001.pdf